CLINICAL TRIAL: NCT03362151
Title: A Clinical Study to Investigate and Compare the Impact of High Protein Pasta, Lower Protein Pasta and White Rice on Blood Sugar Control in People With Type 1 Diabetes Mellitus (T1DM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Harvard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB17-1316
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: type 1 diabetes; pasta; rice; protein; carbohydrate
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Subjects will consume pre-determined meals on 6 difference occasions. There will be three categories of "study meals" consisting of:
  1. Regular pasta (42 grams carbohydrate per meal)
  2. High protein pasta (38 grams carbohydrate per meal)
  3. White rice (43 grams carbohydrate per meal)
  Each subject will consume each meal on two separate occasions in random order.
Who Masked: Participant, Investigator
Masking Description: Subjects will not be told which meal they are eating.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Regular pasta (Experimental): Subjects will bolus rapid acting insulin per their carbohydrate ratio just prior to a meal of regular pasta. They will consume this meal on two separate occasions.
  Interventions: Other: Regular pasta
- High protein pasta (Experimental): Subjects will bolus rapid acting insulin per their carbohydrate ratio just prior to a meal of high protein pasta. They will consume this meal on two separate occasions.
  Interventions: Other: High protein pasta
- White rice (Experimental): Subjects will bolus rapid acting insulin per their carbohydrate ratio just prior to a meal of white rice. They will consume this meal on two separate occasions.
  Interventions: Other: White rice

INTERVENTIONS:
Other: Regular pasta — Regular pasta (Approximately 42 grams carbohydrate per meal)
  Arms: Regular pasta
Other: High protein pasta — High protein pasta (Approximately 38 grams carbohydrate per meal)
  Arms: High protein pasta
Other: White rice — White rice (Approximately 43 grams carbohydrate per meal)
  Arms: White rice

SUMMARY:
The aim of this clinical study is to investigate and compare the postprandial glycemic response to three different meal types rich in carbohydrates, that is, white pasta, high protein pasta and white rice consumed by individuals with T1DM.

DETAILED DESCRIPTION:
The aim of this clinical study is to investigate and compare the postprandial glycemic response to three different meal types rich in carbohydrates, that is, white pasta, high protein pasta and white rice consumed by individuals with T1DM and to demonstrate that:

1. The choice of carbohydrates consumed significantly affects the postprandial glycemic profile in people with type 1 diabetes and
2. The consumption of high protein pasta will present a tighter postprandial glycemic response.

Previous studies have evaluated the effect of white pasta and rice on postprandial glycemic response in people with type 1 diabetes. With this study, we aim to expand upon these findings by ensuring that the results can still be applied to more recent commercial food products (pasta, rice), but especially to evaluate the effect of high-protein pasta when compared to regularly consumed carbohydrates (white pasta, white rice).

After consuming the study meal, subjects will participate in an education session (a 2 hour class per each meal challenge session). Classes will be taught by a registered dietician and diabetes & exercise expert and, as appropriate, a culinary instructor.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75 years at the time of screening.
* Clinical diagnosis of type 1 diabetes for at least one year.
* HbA1c ≤ 10%, as performed by point of care or central laboratory testing. A1c will be assessed at the screening visit, or if already completed within 2 months of the screening visit, the prior lab value may be used in lieu of repeating this assessment.
* Currently using insulin-to-carbohydrate ratio to calculate meal bolus sizes, and boluses for all meals and snacks that contain ≥ 5 grams of carbohydrate.
* Willing to refrain from taking acetaminophen products for the duration of the clinical trial. If acetaminophen is taken, subject is to avoid making any insulin dosing decisions based on CGM for at least 12 hours.
* For females, not currently known to be pregnant. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative urine pregnancy test will be required for all premenopausal women who are not surgically sterile at the screening visit. Subjects who become pregnant will be discontinued from the study.
* Willing to abide by the study protocol and use study-provided devices.

Exclusion Criteria:

* Gastrointestinal disease such as celiac disease or multiple food allergies.
* Any form of gluten sensitivity or wheat allergy.
* Allergies to any form of nuts and ingredients present in the study meals (tomatoes etc).
* History of gastroparesis.
* Pregnancy.
* Dermatological conditions that would preclude wearing a CGM sensor.
* Screening A1c > 10%.
* Any condition that could interfere with participating in the trial, based on the investigator's judgment.
* A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol.
* Participation in another pharmaceutical or device trial at the time of enrollment or during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Delta glucose (maximum rise from baseline glucose) mg/dL | 5 hours
  Delta glucose (maximum rise from baseline glucose) from the start of the meal to the peak continuous glucose monitoring (CGM) glucose reading (mg/dL) during the 5-hour postprandial window, compared between the three meal types.

SECONDARY OUTCOMES:
Incremental area under the curve (area) | 5 hours
  Incremental area under the curve (iAUC) glucose level for the 5 hour postprandial period adjusted for baseline glucose at the start of the meal.
Time to peak glucose level (minutes) | 5 hours
  Time to peak glucose level (in minutes from intervention)
percent time glucose <70 mg/dL | 5 hours
  In case of postprandial hypoglycemia, percent time glucose <70 mg/dL for the 5 hour postprandial period will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: David Eisenberg, MD, Principal Investigator — Harvard School of Public Health (HSPH); Eyal Dassau, PhD, Principal Investigator — Harvard University; Jordan E Pinsker, MD, Principal Investigator — Sansum Diabetes Research Institute
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zavitsanou S, Massa J, Deshpande S, Pinsker JE, Church MM, Andre C, Doyle Iii FJ, Michelson A, Creason J, Dassau E, Eisenberg DM. The Effect of Two Types of Pasta Versus White Rice on Postprandial Blood Glucose Levels in Adults with Type 1 Diabetes: A Randomized Crossover Trial. Diabetes Technol Ther. 2019 Sep;21(9):485-492. doi: 10.1089/dia.2019.0109. Epub 2019 Jun 21. PMID 31225739